CLINICAL TRIAL: NCT04607980
Title: A Phase 3, Multicenter, Randomized, Double-Blind Study Evaluating the Efficacy and Safety of ABP 654 Compared With Ustekinumab in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Investigate ABP 654 for the Treatment of Participants With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20190232; 2020-003184-25 (EudraCT Number)
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; Biosimilar; Psoriasis area and severity index
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigators, study personnel with the exception of the clinical research organization's unblinded biostatistician and unblinded programmers; and the data monitoring committee, and the study participants will remain blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group A (ABP 654) (Experimental): Participants will receive subcutaneous (SC) injection of ABP 654, 45 mg (baseline BW less than equal to [<=] 100 kg) or 90 mg (baseline BW greater than [>] 100 kg) at weeks 0, 4, and 16. Further from week 28 participants will receive ABP 654 (same dose) every 12 weeks (Q12W) at weeks 28 and 40 or may receive dose intensification Q8W at weeks 28, 36, and 44, depending on PASI score.
  Interventions: Drug: ABP 654
- Treatment Group B (Ustekinumab - ABP 654) (Experimental): Participants will receive SC injection of ustekinumab,45 mg (baseline BW <= 100 kg) or 90 mg (baseline BW > 100 kg) at weeks 0, 4, and 16. At week 28, participants will be re-randomized to continue on ustekinumab (Treatment group B1), or to receive ABP 654 (Treatment group B2) on weeks 28 and 40. Depending on PASI score, some participants may not be re-randomized and may receive dose intensification with ustekinumab Q8W at weeks 28, 36, and 44.
  Interventions: Drug: ABP 654; Drug: Ustekinumab

INTERVENTIONS:
Drug: ABP 654 — Participants will receive SC injection of ABP 654.
Drug: Ustekinumab — Participants will receive SC injection of ustekinumab.
  Other Names: Stelara®
  Arms: Treatment Group B (Ustekinumab - ABP 654)

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety, and immunogenicity of ABP 654 compared with ustekinumab in participants with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a multicenter study and will enroll approximately 542 participants.

The total duration of study participation for each participant will be 56 weeks, with up to 4 weeks for screening, and for 52 weeks after the first administration of either ABP 654 or ustekinumab.

After confirmation of eligibility, all participants will be randomized in a 1:1 ratio into 2 treatment groups (Group A will receive ABP 654, and Group B will receive ustekinumab) stratified by prior biologic use for psoriasis (yes versus [vs] no), geographic region, and baseline body weight (BW).

Based on the psoriasis area and severity index (PASI) score (to determine better improvement or partial improvement) at week 28, the participants in the study will proceed as follows:

1. Participants who do not achieve PASI 50 response or better improvement at Week 28 will be considered to have completed the study and will complete end of study procedures (ie, week 52 procedures), and those unable to complete week 28 visit, or did not have a PASI assessment completed, will be discontinued from the study.
2. Participants who achieve PASI 75 response or better improvement will continue on the study and will be re-randomized in a blinded fashion such that participants initially randomized to Group A (ABP 654) will continue to receive ABP 654 and those in Group B (ustekinumab) will re-randomized, to either continue on ustekinumab (Treatment Group B1) or switch to ABP 654 (Treatment Group B2).
3. Participants with PASI 50 response or better but less than PASI 75 response and on the Investigator's decision, participants will continue on the originally assigned treatment with dose intensification and will not be re-randomized. However, participants that do not dose intensify will be re-randomized.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Stable moderate to severe plaque psoriasis for at least 6 months
* Baseline score of PASI >= 12, involvement of >= 10% BSA, and sPGA >= 3 at screening and at baseline
* Candidate for phototherapy or systemic therapy
* Previous failure, inadequate response, intolerance, or contraindication to at least 1 conventional anti-psoriatic systemic therapy
* Female participants should have negative serum pregnancy test during screening and a negative urine pregnancy test at baseline
* No known history of latent or active tuberculosis (TB), and has a negative test for TB during screening (with negative purified protein derivative (PPD), and Negative Quantiferon®/T-spot test)
* Participants with a positive purified protein derivative and a history of Bacillus Calmette-Guérin (BCG) vaccination are allowed with a negative Quantiferon®/T-spot®
* Participants with a positive PPD test (without history of BCG vaccination) or participants with a positive or indeterminate Quantiferon®/T-spot test are allowed if they have all of the following:

  * No symptoms per TB worksheet provided by the sponsor
  * Documented history of adequate prophylaxis initiation prior to receiving investigational product (IP) in accordance with local recommendations
  * No known exposure to a case of active TB after most recent prophylaxis
  * No evidence of active TB on chest radiograph within 3 months prior to the first dose of IP

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Skin disease related conditions such as, Erythrodermic psoriasis (PsO), pustular PsO, guttate PsO, medication induced PsO, or other skin conditions at the time of the screening visit (eg, eczema) that would interfere with evaluations of the effect of IP on PsO
* Participant has an active infection, recurrent or chronic infections, serious infection or history of infections
* Known history of human immunodeficiency virus
* Hepatitis B surface antigen or hepatitis C virus antibody positivity at screening
* Uncontrolled, clinically significant systemic disease such as uncontrolled diabetes mellitus, cardiovascular disease, renal disease, liver disease, or hypertension
* Moderate to severe heart failure (New York Heart Associate class III/IV)
* Known hypersensitivity to the IP or to any of the excipients
* Any abnormal laboratory parameters at screening, as defined in protocol
* Previous treatment with any agent specifically targeting interleukin (IL)-12 or IL-23
* Received biologic treatment for psoriasis within the previous month or 5 drug half-lives prior to randomization
* Received non-biologic systemic psoriasis therapy within 4 weeks prior to randomization
* Received Ultra-violet A (UVA) phototherapy (with or without psoralen) or excimer laser within 4 weeks prior to randomization, or ultra-violet B (UVB) phototherapy within 2 weeks prior to randomization
* Received topical psoriasis treatment within 2 weeks prior to randomization (exception: upper mid-strength to least potent [class III to VII] topical steroids permitted on the palms, soles, face, and intertriginous areas; bland emollients)
* Received live viral or live bacterial vaccination within 2 weeks prior to randomization
* Received BCG vaccination within 1 year prior to randomization
* Other investigational procedures within 4 weeks prior to randomization and during the study
* Participants not agreeing to follow protocol defined contraceptives procedures
* Participants likely not to be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (84):
- United States (34):
  - Total Skin and Beauty Dermatology Center PC, Birmingham, Alabama
  - Alliance Dermatology and Mohs Center, Phoenix, Arizona
  - First OC Dermatology, Fountain Valley, California
  - University Clinical Trials, Inc., San Diego, California
  - San Luis Dermatology and Laser Clinic - Dermatology, San Luis Obispo, California
  - Clinical Science Institute, Santa Monica, California
  - Unison Clinical Trials, Sherman Oaks, California
  - Revival Research, Doral, Florida
  - International Dermatology Research, Inc, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Moore Clinical Research Inc., Tampa, Florida
  - NorthShore University HealthSystem, Skokie, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Epiphany Dermatology of Kansas, LLC, Overland Park, Kansas
  - DelRicht Research, Baton Rouge, Louisiana
  - ALLCUTIS Research, LLC., Beverly, Massachusetts
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - ActivMed Practices & Research, LLC., Portsmouth, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Dermatology Consulting Services, PLLC, High Point, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - Dermatologists of Southwest Ohio, Mason, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - The Pennsylvania Centre for Dermatology, LLC, Exton, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - The Skin Wellness Center PC, Knoxville, Tennessee
  - Center for Clinical Studies, Cypress, Texas
  - Modern Research Associates, Dallas, Texas
  - Austin Institute for Clinical Research - Dermatology, Houston, Texas
  - Progressive Clinical Research [Texas], San Antonio, Texas
  - Acclaim Dermatology, Sugar Land, Texas
- Canada (15):
  - Beacon Dermatology, Calgary, Alberta
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - CCA Medical Research, Ajax, Ontario
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Dermatrials Research Inc, Hamilton, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - DermEdge Research Inc., Mississauga, Ontario
  - North Bay Dermatology Centre Inc., North Bay, Ontario
  - JRB Research Inc., Ottawa, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - Toronto Research Centre - Dermatology, Toronto, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
  - XLR8 Medical Research Inc., Windsor, Ontario
  - Centre de Recherche dermatolog, Québec, Quebec
- Estonia (4):
  - Vahlberg & Pild OÜ, Tallinn, Harju
  - Confido Private Medical Clinic - General Practice/Medicine, Tallinn, Harju
  - Clinical Research Center, Tartu, Tartu
  - Tartu University Hospital, Tartu, Tartu
- Germany (4):
  - Dermatologische Gemeinschaftspraxis Dres.Scholz Sebastian Schilling, Mahlow, Brandenburg
  - Derma Zentrum Osnabrueck Nord, Bramsche, Lower Saxony
  - Hautzentrum im Jahrhunderthaus, Bochum, North Rhine-Westphalia
  - CentroDerm GmbH, Wuppertal, North Rhine-Westphalia
- Hungary (2):
  - Brgyógyászati és Allergológiai Magánrendelés, Szolnok, Jász-Nagykun-Szolnok
  - UNOMEDICALTRIALS Kft, Budapest, Pest County
- Latvia (5):
  - Health Centre 4 Ltd., Diagnostics Centre, Riga, Rga
  - Riga 1st hospital, Clinic of Dermatology and STD, Riga, Rga
  - J.Kisis LtD, Riga, Rga
  - Health and Aesthetics Ltd, Riga
  - Smite Aija doctor practice in dermatology, venereology, Talsi
- Lithuania (2):
  - Lietuvos sveikatos mokslu universiteto ligonine Kauno klinik, Kaunas, Kaunas County
  - Vilniaus universiteto ligonine Santaros klinikos Dermatovenerologijos centras, Vilnius, Vilnius County
- Poland (18):
  - Centrum Medyczne ALL-MED, Krakow, Maopolskie
  - Medycyna Kliniczna, Warsaw, Masovian Voivodeship
  - ETG Warszawa, Warsaw, Masovian Voivodeship
  - Royalderm Agnieszka Nawrocka, Warsaw, Masovian Voivodeship
  - Zespol Naukowo-Leczniczy Iwolang sp. z.o.o., Iwonicz-Zdrój, Podkarpackie Voivodeship
  - Specderm Poznanska Sp. j., Bialystok, Podlaskie Voivodeship
  - ClinicMed Daniluk, Nowak Sp. J., Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Pratia Katowice, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Barbara Rewerska Diamond Clinic, Krakow
  - Centrum Zdrowia i Urody Maxxmed, Lublin
  - ETG Lublin, Lublin
  - Solumed, Poznan
  - Nasz Lekarz Osrodek Badan Klinicznych, Torun
  - Klinika Ambroziak Dermatologia, Warsaw
  - DermMedica Sp. z o.o., Wroclaw
  - WroMedica I. Bielicka, A. Strzalkowska s.c., Wroclaw
  - ETG Skierniewice, Skierniewice, Ódzkie

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Blauvelt A, Papp K, Trivedi M, Barragan C, Chow V, Mytych DT, Yamauchi P, Crowley J, Franklin J. Efficacy and safety of the ustekinumab biosimilar ABP 654 in patients with moderate-to-severe plaque psoriasis: a randomized double-blinded active-controlled comparative clinical study over 52 weeks. Br J Dermatol. 2025 Apr 28;192(5):826-836. doi: 10.1093/bjd/ljae402. PMID 39442018
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 84 centers in Canada, Estonia, Germany, Hungary, Latvia, Lithuania, Poland, and the United States between 11 November 2020 and 03 June 2022.
Pre-assignment Details: Of the 648 participants screened, 563 participants were enrolled and randomized in a 1:1 ratio to receive ABP 654 or ustekinumab.
Groups:
- Treatment Group A (ABP 654): Participants received SC injection of ABP 654, 45 mg (Baseline body weight [BW] less than or equal to [<=] 100 kg) or 90 mg (Baseline BW greater than [>] 100 kg) at Weeks 0, 4, and 16. From Week 28 participants received ABP 654 (same dose) every 12 weeks (Q12W) at Weeks 28 and 40 or depending on Psoriasis Area and Severity Index (PASI) score, received dose intensification every 8 weeks (Q8W) at Weeks 28, 36, and 44 (as per protocol).
- Treatment Group B (Ustekinumab): Participants received SC injection of ustekinumab, 45 mg (Baseline BW <= 100 kg) or 90 mg (Baseline BW > 100 kg) at Weeks 0, 4, and 16. At Week 28, participants were re-randomized to continue receiving ustekinumab (Treatment group B1), or to receive ABP 654 (Treatment group B2) at Weeks 28 and 40. Depending on PASI score, some participants were not re-randomized and received dose intensification with ustekinumab Q8W at Weeks 28, 36, and 44 (as per protocol).
Period: Overall Study
Arm/Group | Treatment Group A (ABP 654) | Treatment Group B (Ustekinumab)
Started | 281 | 282
Treated | 280 | 282
Re-randomized to ABP 654 at Week 28 | 247 | 117
Re-randomized to Ustekinumab at Week 28 | 0 | 116
Not Re-randomized at Week 28 and Dose Intensified | 25 | 34
Completed | 269 | 261
Not Completed | 12 | 21
Not completed — Adverse Event | 3 | 4
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Lost to Follow-up | 4 | 8
Not completed — Protocol Violation | 0 | 3
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): consisted of all randomized participants.
Groups:
- Treatment Group A (ABP 654): Participants received SC injection of ABP 654, 45 mg (Baseline BW <= 100 kg) or 90 mg (Baseline BW > 100 kg) at Weeks 0, 4, and 16. From Week 28 participants received ABP 654 (same dose) Q12W at Weeks 28 and 40 or, depending on PASI score, received dose intensification Q8W at Weeks 28, 36, and 44 (as per protocol).
- Total: Total of all reporting groups
Arm/Group | Treatment Group A (ABP 654) | Treatment Group B (Ustekinumab) | Total
Number analyzed (Participants) | 281 | 282 | 563
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (14.15) | 45.0 (12.58) | 44.4 (13.39)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 257 | 261 | 518
  From 65-84 years | 24 | 21 | 45
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 91 | 195
  Male | 177 | 191 | 368
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 20 | 25 | 45
  Black or African American | 4 | 2 | 6
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White | 250 | 247 | 497
  Multiple | 1 | 0 | 1
  Not allowed to collect | 1 | 0 | 1
  Other | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 28 | 60
  Not Hispanic or Latino | 248 | 252 | 500
  Not allowed to collect | 1 | 0 | 1
  Unknown | 0 | 2 | 2
Static Physician Global Assessment of Psoriasis (sPGA) [Count of Participants; unit: Participants] — The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema).
  Participants
    Score 0 (clear) | 0 | 0 | 0
    Score 1 (almost clear) | 0 | 0 | 0
    Score 2 (mild) | 0 | 0 | 0
    Score 3 (moderate) | 130 | 154 | 284
    Score 4 (severe) | 132 | 114 | 246
    Score 5 (very severe) | 19 | 14 | 33
PASI [Mean (Standard Deviation); unit: Score on a scale] — The PASI is a measure of the average redness (erythema), thickness (induration), and scaliness (scaling; each graded on a 0-4 scale [0 = clear; 1-4 = increasing severity]) of the lesions, weighted by the area of involvement in the four main body areas (i.e., head, arms, trunk to groin, and legs to top of buttocks). The PASI score ranges from 0 to 72. Higher scores represent worse symptom severity.
  Score on a scale | 21.50 (8.855) | 20.35 (7.850) | 20.92 (8.379)
Psoriasis Body Surface Area (BSA) [Mean (Standard Deviation); unit: Percentage of BSA] — The percentage of BSA affected was estimated by assuming that the participant's palm, excluding the fingers and thumb, represents roughly 1% of the body's surface.
  Percentage of BSA | 26.5 (15.25) | 24.9 (15.05) | 25.7 (15.16)

OUTCOME MEASURES:

1. Primary Outcome: PASI Percent Change From Baseline to Week 12
Description: The PASI is a measure of the average redness (erythema), thickness (induration), and scaliness (scaling; each graded on a 0-4 scale [0 = clear; 1-4 = increasing severity]) of the lesions, weighted by the area of involvement in the four main body areas (i.e., head, arms, trunk to groin, and legs to top of buttocks). The PASI score ranges from 0 to 72. Higher scores represent worse symptom severity.
Time Frame: Baseline (Day 1 [Week 0]) and Week 12
Population: Results are presented for the FAS with available data; observed data was used for summary statistics.
Measure: Mean (Standard Deviation); unit: Percent Change in PASI score
Arm/Group | Treatment Group A (ABP 654) | Treatment Group B (Ustekinumab)
Number analyzed (Participants) | 272 | 276
Percent Change in PASI score | 81.92 (19.872) [lower limit 19.872] | 81.91 (19.611) [lower limit 19.611]
Statistical Analysis 1: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Multiple imputation was applied for the point estimate and CI of the mean difference between the 2 groups; Test type: Equivalence — Clinical equivalence of the primary endpoint was evaluated by comparing the 2-sided 95% confidence interval (CI) of the mean difference of PASI percent improvement from Baseline to Week 12 between ABP 654 versus (vs) ustekinumab with an equivalence margin of (-15, +15); Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-3.16 to 3.43]

2. Secondary Outcome: PASI Percent Change at Other Timepoints
Description: as for outcome 1
Time Frame: Baseline (Day 1 [Week 0]), Weeks 4, 16, 28, 36 (dose intensification only), 40 (re-randomized FAS only), 44 (dose intensification only) and Week 52 (End of Study [EOS])
Population: Through Week 28 results are presented for the FAS with available data; last observation carried forward (LOCF) imputation was used. Post Week 28 results are presented for dose intensification participants with available observed data and re-randomized FAS participants with available data (LOCF imputation was used).
Measure: Mean (Standard Deviation); unit: Percent Change in PASI score
Groups:
- Post Week 28: ABP 654/ ABP 654: All participants who were randomized to receive SC injection of ABP 654 at Weeks 0, 4, and 16, followed by ABP 654 (same dose) Q12W at Weeks 28 and 40.
- Post Week 28: Ustekinumab/ ABP 654: All participants who were randomized to receive SC injection of ustekinumab at Weeks 0, 4, and 16. At Week 28, participants were re-randomized to receive ABP 654 (Treatment group B2) at Weeks 28 and 40.
- Post Week 28: Ustekinumab/ Ustekinumab: All participants who were randomized to receive SC injection of ustekinumab at Weeks 0, 4, and 16. At Week 28, participants were re-randomized to continue on ustekinumab (Treatment group B1) at Weeks 28 and 40.
Arm/Group | Treatment Group A (ABP 654) | Treatment Group B (Ustekinumab) | Post Week 28: ABP 654/ ABP 654 | Post Week 28: Ustekinumab/ ABP 654 | Post Week 28: Ustekinumab/ Ustekinumab
Number analyzed (Participants) | 280 | 281 | 247 | 117 | 116
Percent Change in PASI score
  Week 4: number analyzed (Participants) | 280 | 281 | 0 | 0 | 0
  Week 4 | 44.15 (23.587) | 42.40 (24.536) |  |  |
  Week 16: number analyzed (Participants) | 280 | 281 | 0 | 0 | 0
  Week 16 | 85.88 (18.704) | 85.86 (19.953) |  |  |
  Week 28: number analyzed (Participants) | 280 | 281 | 0 | 0 | 0
  Week 28 | 89.41 (14.228) | 88.18 (18.771) |  |  |
  Week 36: number analyzed (Participants) | 25 | 34 | 0 | 0 | 0
  Week 36 | 75.53 (11.038) | 74.12 (13.826) |  |  |
  Week 40: number analyzed (Participants) | 0 | 0 | 247 | 117 | 116
  Week 40 |  |  | 93.60 (9.738) | 94.22 (8.296) | 95.10 (8.529)
  Week 44: number analyzed (Participants) | 25 | 34 | 0 | 0 | 0
  Week 44 | 75.33 (15.563) | 78.42 (14.733) |  |  |
  Week 52: number analyzed (Participants) | 25 | 34 | 247 | 117 | 116
  Week 52 | 77.80 (14.760) | 77.46 (18.109) | 92.54 (11.808) | 93.90 (8.987) | 93.23 (16.029)
Statistical Analysis 1: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 4: Treatment Group A vs Treatment Group B. LOCF imputation was used; Test type: Equivalence — The mean differences and 95% CIs of PASI percent improvement between the initial randomized groups (ABP 654 vs ustekinumab) at other scheduled visits was estimated using analysis of covariance (ANCOVA) model adjusted for baseline PASI value, and the stratification factors of prior biologic use for psoriasis, baseline BW group, and geographic region; Mean Difference (Final Values) = 1.95, 95% CI 2-sided [-2.05 to 5.94]
Statistical Analysis 2: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 16: Treatment Group A vs Treatment Group B. LOCF imputation was used; Test type: Equivalence — The mean differences and 95% CIs of PASI percent improvement between the initial randomized groups (ABP 654 vs ustekinumab) at other scheduled visits was estimated using ANCOVA model adjusted for baseline PASI value, and the stratification factors of prior biologic use for psoriasis, baseline BW group, and geographic region; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-2.97 to 3.31]
Statistical Analysis 3: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 28: Treatment Group A vs Treatment Group B. LOCF imputation was used; Test type: Equivalence — [test comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = 1.34, 95% CI 2-sided [-1.39 to 4.07]
Statistical Analysis 4: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 36: Treatment Group A vs Treatment Group B. Observed data was used; Test type: Equivalence — The mean differences and 95% CIs of PASI percent improvement between the dose intensification groups (ABP 654 vs ustekinumab) at other scheduled visits was estimated using ANCOVA model adjusted for baseline PASI value, and the stratification factors of prior biologic use for psoriasis, baseline BW group, and geographic region; Mean Difference (Final Values) = 1.26, 95% CI 2-sided [-5.46 to 7.98]
Statistical Analysis 5: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 44: Treatment Group A vs Treatment Group B. Observed data was used; Test type: Equivalence — [test comment as in outcome 2, analysis 4]; Mean Difference (Final Values) = -3.71, 95% CI 2-sided [-10.71 to 3.28]
Statistical Analysis 6: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 52: Treatment Group A vs Treatment Group B. Observed data was used; Test type: Equivalence — [test comment as in outcome 2, analysis 4]; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-8.45 to 7.13]
Statistical Analysis 7: Comparison: Post Week 28: ABP 654/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 40: ABP 654 vs Ustekinumab. LOCF imputation was used; Test type: Equivalence — The differences for the mean percent change from baseline and the corresponding CIs were for ABP 654/ABP 654 minus ustekinumab/ustekinumab. Estimated using ANCOVA model adjusted for baseline PASI value, and the stratification factors of prior biologic use for psoriasis, baseline BW group, and geographic region; Mean Difference (Final Values) = -1.41, 95% CI 2-sided [-3.42 to 0.59]
Statistical Analysis 8: Comparison: Post Week 28: Ustekinumab/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 40: Ustekinumab/ABP 654 vs Ustekinumab. LOCF imputation was used; Test type: Equivalence — The differences for the mean percent change from baseline and the corresponding CIs were for ustekinumab/ABP 654 minus ustekinumab/ustekinumab. Estimated using ANCOVA model adjusted for baseline PASI value, and the stratification factors of prior biologic use for psoriasis, baseline BW group, and geographic region; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-3.17 to 1.48]
Statistical Analysis 9: Comparison: Post Week 28: ABP 654/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 52: ABP 654 vs Ustekinumab. LOCF imputation was used; Test type: Equivalence — [test comment as in outcome 2, analysis 7]; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-3.29 to 2.17]
Statistical Analysis 10: Comparison: Post Week 28: Ustekinumab/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 52: Ustekinumab/ABP 654 vs Ustekinumab. LOCF imputation was used; Test type: Equivalence — [test comment as in outcome 2, analysis 8]; Mean Difference (Final Values) = 0.70, 95% CI 2-sided [-2.46 to 3.86]

3. Secondary Outcome: Percentage of Participants With PASI 75 Response Throughout the Study
Description: Reduction in disease was measured by PASI score. The PASI 75 response is a 75% or greater improvement (reduction in disease [PASI 75]) from baseline in PASI score. The PASI is a measure of the average redness (erythema), thickness (induration), and scaliness (scaling; each graded on a 0-4 scale [0 = clear; 1-4 = increasing severity]) of the lesions, weighted by the area of involvement in the four main body areas (i.e., head, arms, trunk to groin, and legs to top of buttocks). The PASI score ranges from 0 to 72. Higher scores represent worse symptom severity.
Time Frame: Baseline (Day 1 [Week 0]), Weeks 4, 16, 28, 36 (dose intensification only), 40 (re-randomized FAS only), 44 (dose intensification only) and Week 52 (EOS)
Population: Through Week 28 FAS results are presented for the FAS with available data; non-responder imputation (NRI) was used. Post Week 28 results are presented for dose intensification participants with available observed data and re-randomized FAS participants with available data (NRI was used).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment Group A (ABP 654) | Treatment Group B (Ustekinumab) | Post Week 28: ABP 654/ ABP 654 | Post Week 28: Ustekinumab/ ABP 654 | Post Week 28: Ustekinumab/ Ustekinumab
Number analyzed (Participants) | 281 | 282 | 247 | 117 | 116
Percentage of participants
  Week 4: number analyzed (Participants) | 281 | 282 | 0 | 0 | 0
  Week 4 | 11.4 [7.67 to 15.10] | 10.3 [6.74 to 13.83] |  |  |
  Week 12: number analyzed (Participants) | 281 | 282 | 0 | 0 | 0
  Week 12 | 69.8 [64.38 to 75.12] | 70.2 [64.88 to 75.55] |  |  |
  Week 16: number analyzed (Participants) | 281 | 282 | 0 | 0 | 0
  Week 16 | 80.8 [76.18 to 85.39] | 80.1 [75.49 to 84.80] |  |  |
  Week 28: number analyzed (Participants) | 281 | 282 | 0 | 0 | 0
  Week 28 | 85.8 [81.68 to 89.85] | 82.3 [77.81 to 86.73] |  |  |
  Week 36: number analyzed (Participants) | 25 | 34 | 0 | 0 | 0
  Week 36 | 52.0 [32.42 to 71.58] | 55.9 [39.19 to 72.57] |  |  |
  Week 40: number analyzed (Participants) | 0 | 0 | 247 | 117 | 116
  Week 40 |  |  | 94.7 [91.95 to 97.52] | 95.7 [92.06 to 99.39] | 94.0 [89.63 to 98.30]
  Week 44: number analyzed (Participants) | 25 | 34 | 0 | 0 | 0
  Week 44 | 48.0 [28.42 to 67.58] | 64.7 [48.64 to 80.77] |  |  |
  Week 52: number analyzed (Participants) | 25 | 34 | 247 | 117 | 116
  Week 52 | 64.0 [45.18 to 82.82] | 58.8 [42.28 to 75.37] | 89.5 [85.65 to 93.30] | 92.3 [87.48 to 97.14] | 92.2 [87.37 to 97.11]
Statistical Analysis 1: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 4: Treatment Group A vs Treatment Group B. NRI was used; Test type: Equivalence — Response difference (ABP 654 - ustekinumab) was estimated by the Mantel-Haenszel estimate, and the 95% CIs were estimated by the stratified Newcombe confidence limits, adjusting for actual stratification factors of prior biologic use for psoriasis, baseline BW group, and geographic region; Response difference = 1.20, 95% CI 2-sided [-4.02 to 6.42]
Statistical Analysis 2: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 12: Treatment Group A vs Treatment Group B. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Response difference = -0.32, 95% CI 2-sided [-7.87 to 7.23]
Statistical Analysis 3: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 16: Treatment Group A vs Treatment Group B. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Response difference = 0.82, 95% CI 2-sided [-5.75 to 7.37]
Statistical Analysis 4: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 28: Treatment Group A vs Treatment Group B. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Response difference = 3.75, 95% CI 2-sided [-2.37 to 9.84]
Statistical Analysis 5: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 36: Treatment Group A vs Treatment Group B. Observed data was used; Test type: Equivalence — Response difference in dose intensification participants (ABP 654 - ustekinumab) was estimated by the generalized linear model adjusted for the baseline PASI and the stratification factors with an identity link was used to obtain the point estimate and 95% CI for the risk difference of PASI 75 response rate at each scheduled timepoint; Response difference = -3.19, 95% CI 2-sided [-28.15 to 21.76]
Statistical Analysis 6: Comparison: Post Week 28: ABP 654/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 40: ABP 654 vs Ustekinumab. NRI was used; Test type: Equivalence — Response difference (ABP 654/ABP 654 - ustekinumab/ustekinumab) was estimated by the Mantel-Haenszel estimate, and the 95% CIs were estimated by the stratified Newcombe confidence limits, adjusting for actual stratification factors of prior biologic use for psoriasis, baseline BW group, and geographic region; Response difference = 1.10, 95% CI 2-sided [-3.74 to 7.54]
Statistical Analysis 7: Comparison: Post Week 28: Ustekinumab/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 40: Ustekinumab/ABP 654 vs Ustekinumab. NRI was used; Test type: Equivalence — Response difference (ustekinumab/ABP 654 - ustekinumab/ustekinumab) was estimated by the Mantel-Haenszel estimate, and the 95% CIs were estimated by the stratified Newcombe confidence limits, adjusting for actual stratification factors of prior biologic use for psoriasis, baseline BW group, and geographic region; Response difference = 1.85, 95% CI 2-sided [-4.89 to 8.39]
Statistical Analysis 8: Comparison: Post Week 28: ABP 654/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 52: ABP 654 vs Ustekinumab. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 6]; Response difference = -2.75, 95% CI 2-sided [-8.61 to 4.41]
Statistical Analysis 9: Comparison: Post Week 28: Ustekinumab/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 52: Ustekinumab/ABP 654 vs Ustekinumab. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 7]; Response difference = 0.14, 95% CI 2-sided [-7.32 to 7.43]

4. Secondary Outcome: Percentage of Participants With PASI 100 Response Throughout the Study
Description: Reduction in disease was measured by PASI score. The PASI 100 response is a 100% improvement (reduction in disease [PASI 100]) from baseline in PASI score. The PASI is a measure of the average redness (erythema), thickness (induration), and scaliness (scaling; each graded on a 0-4 scale [0 = clear; 1-4 = increasing severity]) of the lesions, weighted by the area of involvement in the four main body areas (i.e., head, arms, trunk to groin, and legs to top of buttocks). The PASI score ranges from 0 to 72. Higher scores represent worse symptom severity.
Time Frame: as for outcome 3
Population: Through Week 28 FAS results are presented for the FAS with available data; NRI was used. Post Week 28 results are presented for dose intensification participants with available observed data and re-randomized FAS participants with available data (NRI was used).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment Group A (ABP 654) | Treatment Group B (Ustekinumab) | Post Week 28: ABP 654/ ABP 654 | Post Week 28: Ustekinumab/ ABP 654 | Post Week 28: Ustekinumab/ Ustekinumab
Number analyzed (Participants) | 281 | 282 | 247 | 117 | 116
Percentage of participants
  Week 4: number analyzed (Participants) | 281 | 282 | 0 | 0 | 0
  Week 4 | 0.4 [0.00 to 1.05] | 0.7 [0.00 to 1.69] |  |  |
  Week 12: number analyzed (Participants) | 281 | 282 | 0 | 0 | 0
  Week 12 | 20.6 [15.91 to 25.37] | 19.1 [14.56 to 23.74] |  |  |
  Week 16: number analyzed (Participants) | 281 | 282 | 0 | 0 | 0
  Week 16 | 29.9 [24.54 to 35.25] | 26.2 [21.11 to 31.38] |  |  |
  Week 28: number analyzed (Participants) | 281 | 282 | 0 | 0 | 0
  Week 28 | 34.5 [28.96 to 40.08] | 31.6 [26.14 to 36.98] |  |  |
  Week 36: number analyzed (Participants) | 25 | 34 | 0 | 0 | 0
  Week 36 | 0 [NA to NA] — CIs were not estimable as there were no PASI responses. | 0 [NA to NA] — CIs were not estimable as there were no PASI responses. |  |  |
  Week 40: number analyzed (Participants) | 0 | 0 | 247 | 117 | 116
  Week 40 |  |  | 44.5 [38.34 to 50.73] | 41.9 [32.94 to 50.82] | 46.6 [37.47 to 55.63]
  Week 44: number analyzed (Participants) | 25 | 34 | 0 | 0 | 0
  Week 44 | 4.0 [0.00 to 11.68] | 2.9 [0.00 to 8.62] |  |  |
  Week 52: number analyzed (Participants) | 25 | 34 | 247 | 117 | 116
  Week 52 | 4.0 [0.00 to 11.68] | 14.7 [2.80 to 26.61] | 47.0 [40.74 to 53.19] | 42.7 [33.77 to 51.70] | 44.8 [35.78 to 53.88]
Statistical Analysis 1: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 4: Treatment Group A vs Treatment Group B. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Response difference = -0.34, 95% CI 2-sided [-3.16 to 3.21]
Statistical Analysis 2: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 12: Treatment Group A vs Treatment Group B. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Response difference = 1.58, 95% CI 2-sided [-5.03 to 8.18]
Statistical Analysis 3: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 16: Treatment Group A vs Treatment Group B. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Response difference = 3.81, 95% CI 2-sided [-3.62 to 11.17]
Statistical Analysis 4: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 28: Treatment Group A vs Treatment Group B. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Response difference = 3.07, 95% CI 2-sided [-4.68 to 10.78]
Statistical Analysis 5: Comparison: Post Week 28: ABP 654/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 40: ABP 654 vs Ustekinumab. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 6]; Response difference = -1.93, 95% CI 2-sided [-12.85 to 8.89]
Statistical Analysis 6: Comparison: Post Week 28: Ustekinumab/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 40: Ustekinumab/ABP 654 vs Ustekinumab. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 7]; Response difference = -4.93, 95% CI 2-sided [-17.39 to 7.73]
Statistical Analysis 7: Comparison: Post Week 28: ABP 654/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 52: ABP 654 vs Ustekinumab. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 6]; Response difference = 2.55, 95% CI 2-sided [-8.42 to 13.30]
Statistical Analysis 8: Comparison: Post Week 28: Ustekinumab/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 52: Ustekinumab/ABP 654 vs Ustekinumab. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 7]; Response difference = -2.41, 95% CI 2-sided [-14.91 to 10.19]

5. Secondary Outcome: Percentage of Participants With sPGA Responses (0/1) at Week 12 and Week 52
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). A sPGA response was defined as a sPGA value of clear (score 0) or almost clear (score 1). Higher scores represent worse symptom severity.
Time Frame: Week 12 and Week 52 (EOS)
Population: Week 12 results are presented for the FAS with available data; NRI was used. Week 52 results are presented for dose intensification participants with available data and re-randomized FAS participants with available data (NRI was used).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment Group A (ABP 654) | Treatment Group B (Ustekinumab) | Post Week 28: ABP 654/ ABP 654 | Post Week 28: Ustekinumab/ ABP 654 | Post Week 28: Ustekinumab/ Ustekinumab
Number analyzed (Participants) | 281 | 282 | 247 | 117 | 116
Percentage of participants
  Week 12: number analyzed (Participants) | 281 | 282 | 0 | 0 | 0
  Week 12 | 55.2 [49.35 to 60.98] | 52.8 [47.01 to 58.66] |  |  |
  Week 52: number analyzed (Participants) | 25 | 34 | 247 | 117 | 116
  Week 52 | 24.0 [7.26 to 40.74] | 35.3 [19.23 to 51.36] | 71.3 [65.61 to 76.90] | 70.9 [62.71 to 79.17] | 78.4 [70.97 to 85.93]
Statistical Analysis 1: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 12: Treatment Group A vs Treatment Group B. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Response difference = 2.55, 95% CI 2-sided [-5.65 to 10.71]
Statistical Analysis 2: Comparison: Post Week 28: ABP 654/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 52: ABP 654 vs Ustekinumab. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 6]; Response difference = -6.57, 95% CI 2-sided [-15.41 to 3.29]
Statistical Analysis 3: Comparison: Post Week 28: Ustekinumab/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 52: ABP 654/Ustekinumab vs Ustekinumab. NRI was used; Test type: Equivalence — [test comment as in outcome 3, analysis 7]; Response difference = -7.46, 95% CI 2-sided [-18.41 to 3.74]

6. Secondary Outcome: Change From Baseline in Percentage of BSA Affected With Psoriasis at Week 12 and Week 52
Description: The percentage of BSA affected was estimated by assuming that the participant's palm, excluding the fingers and thumb, represents roughly 1% of the body's surface.
Time Frame: Baseline (Day 1 [Week 0]), Week 12 and Week 52 (EOS)
Population: Week 12 results are presented for the FAS with available data; LOCF imputation was used. Week 52 results are presented for dose intensification participants with available observed data and re-randomized FAS participants with available data (LOCF imputation was used).
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | Treatment Group A (ABP 654) | Treatment Group B (Ustekinumab) | Post Week 28: ABP 654/ ABP 654 | Post Week 28: Ustekinumab/ ABP 654 | Post Week 28: Ustekinumab/ Ustekinumab
Number analyzed (Participants) | 280 | 281 | 247 | 117 | 116
Percentage of BSA
  Week 12: number analyzed (Participants) | 280 | 281 | 0 | 0 | 0
  Week 12 | -17.8 (14.32) | -17.2 (14.51) |  |  |
  Week 52: number analyzed (Participants) | 25 | 34 | 247 | 117 | 116
  Week 52 | -20.6 (14.72) | -21.6 (16.89) | -24.7 (14.81) | -22.8 (13.86) | -22.5 (14.11)
Statistical Analysis 1: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 12: Treatment Group A vs Treatment Group B. LOCF imputation was used; Test type: Equivalence — Mean difference estimated for treatment group A and treatment group B using ANCOVA model adjusted for baseline BSA value, and the stratification factors of prior biologic use for psoriasis, baseline BW group, and geographic region; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-1.15 to 2.10]
Statistical Analysis 2: Comparison: Treatment Group A (ABP 654) vs Treatment Group B (Ustekinumab); Week 52: Treatment Group A vs Treatment Group B. Observed data was used; Test type: Equivalence — Mean difference estimated in dose intensification participants (treatment group A and treatment group B) using ANCOVA model adjusted for baseline BSA value, and the stratification factors of prior biologic use for psoriasis, baseline BW group, and geographic region; Mean Difference (Final Values) = 1.39, 95% CI 2-sided [-0.90 to 3.67]
Statistical Analysis 3: Comparison: Post Week 28: ABP 654/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 52: ABP 654 vs Ustekinumab. LOCF imputation was used; Test type: Equivalence — Mean difference estimated for ABP 654/ ABP 654 and ustekinumab/ ustekinumab using ANCOVA model adjusted for baseline BSA value, and the stratification factors of prior biologic use for psoriasis, baseline BW group, and geographic region; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.99 to 0.74]
Statistical Analysis 4: Comparison: Post Week 28: Ustekinumab/ ABP 654 vs Post Week 28: Ustekinumab/ Ustekinumab; Week 52: Ustekinumab/ABP 654 vs Ustekinumab. LOCF imputation was used; Test type: Equivalence — Mean difference estimated for ustekinumab/ABP 654 and ustekinumab/ ustekinumab using ANCOVA model adjusted for baseline BSA value, and the stratification factors of prior biologic use for psoriasis, baseline BW group, and geographic region; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.90 to 1.10]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were summarized by actual treatment received. For each category, participants were included only once, even if they experienced multiple events in that category.
Time Frame: Day 1 (Week 0) to Week 28; Week 28 to Week 52 (EOS)
Population: Through Week 28 results are presented for the Safety Analysis Set. Post Week 28 results are presented for the re-randomized Safety Analysis Set and the dose intensification participants.
Measure: Count of Participants; unit: Participants
Groups:
- Through Week 28: ABP 654: All participants who were randomized to receive SC injection of ABP 654, 45 mg (Baseline BW <= 100 kg) or 90 mg (Baseline BW > 100 kg) at Weeks 0, 4, and 16.
- Through Week 28: Ustekinumab: All participants who were randomized to receive SC injection of ustekinumab, 45 mg (Baseline BW <= 100 kg) or 90 mg (Baseline BW > 100 kg) at Weeks 0, 4, and 16.
- Post Week 28: ABP 654 Dose Intensification: All participants who were randomized to receive SC injection of ABP 654 at Weeks 0, 4, and 16 with PASI 50 response or better but less than PASI 75 response at Week 28 (as per protocol). Based on the Investigator's discretion, the participants received ABP 654 dose intensification Q8W at Weeks 28, 36, and 44.
- Post Week 28: Ustekinumab Dose Intensification: All participants who were randomized to receive SC injection of ustekinumab at Weeks 0, 4, and 16 with PASI 50 response or better but less than PASI 75 response at Week 28 (as per protocol). Based on the Investigator's discretion, the participants received ustekinumab dose intensification Q8W at Weeks 28, 36, and 44.
Arm/Group | Through Week 28: ABP 654 | Through Week 28: Ustekinumab | Post Week 28: ABP 654/ ABP 654 | Post Week 28: Ustekinumab/ ABP 654 | Post Week 28: Ustekinumab/ Ustekinumab | Post Week 28: ABP 654 Dose Intensification | Post Week 28: Ustekinumab Dose Intensification
Number analyzed (Participants) | 280 | 282 | 247 | 117 | 116 | 25 | 34
Participants
  Any TEAE | 106 | 99 | 85 | 44 | 40 | 12 | 9
  Any Serious TEAE | 7 | 5 | 1 | 1 | 3 | 1 | 0

8. Secondary Outcome: Number of Participants With Events of Interests (EOIs)
Description: The EOIs pre-specified for this study included serious systemic hypersensitivity reactions, facial palsy, pustular psoriasis, erythrodermic psoriasis, serious infections (including mycobacterial and salmonella infections), malignancy, cardiovascular events, reversible posterior leukoencephalopathy syndrome, serious depression including suicidality, and venous thromboembolism.
Time Frame: Day 1 (Week 0) to Week 28; Week 28 to Week 52 (EOS)
Population: Through Week 28 results are presented for the Safety Analysis Set. Post Week 28 results are presented for the re-randomized Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Through Week 28: ABP 654 | Through Week 28: Ustekinumab | Post Week 28: ABP 654/ ABP 654 | Post Week 28: Ustekinumab/ ABP 654 | Post Week 28: Ustekinumab/ Ustekinumab
Number analyzed (Participants) | 280 | 282 | 247 | 117 | 116
Participants | 5 | 7 | 3 | 0 | 4

9. Secondary Outcome: Number of Participants Developing Anti-drug Antibodies (ADAs) to ABP 654
Description: A participant was considered to have developed ADAs if they:
  * had a positive post-baseline binding or neutralizing antibody result with a negative or no result at Baseline or
  * had a positive post-baseline binding or neutralizing antibody result with a negative or no result prior to the first dose in the post Week 28 study period.
Time Frame: Baseline; Day 1 (Week 0) to Week 28; Week 28 to Week 52 (EOS)
Population: Through Week 28 results are presented for the Safety Analysis Set with available ADA data. Post Week 28 results are presented for the re-randomized Safety Analysis Set and dose intensification participants with available ADA data.
Measure: Count of Participants; unit: Participants
Arm/Group | Through Week 28: ABP 654 | Through Week 28: Ustekinumab | Post Week 28: ABP 654/ ABP 654 | Post Week 28: Ustekinumab/ ABP 654 | Post Week 28: Ustekinumab/ Ustekinumab | Post Week 28: ABP 654 Dose Intensification | Post Week 28: Ustekinumab Dose Intensification
Number analyzed (Participants) | 279 | 280 | 246 | 116 | 115 | 25 | 34
Participants
  Binding antibody | 52 | 104 | 11 | 4 | 2 | 0 | 2
  Neutralizing antibody | 24 | 50 | 5 | 1 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 (Week 0) to Week 28; Week 28 to Week 52 (EOS)
Description: Through Week 28: Safety Analysis Set. Post Week 28: Re-randomized Safety Analysis Set.
Groups:
- Post Week 28: ABP 654 / ABP 654: All participants who were randomized to receive SC injection of ABP 654 at Weeks 0, 4, and 16, followed by ABP 654 (same dose) Q12W at Weeks 28 and 40.
- Post Week 28: Ustekinumab / ABP654: All participants who were randomized to receive SC injection of ustekinumab at Weeks 0, 4, and 16. At Week 28, participants were re-randomized to receive ABP 654 (Treatment group B2) at Weeks 28 and 40.
- Post Week 28: Ustekinumab / Ustekinumab: All participants who were randomized to receive SC injection of ustekinumab at Weeks 0, 4, and 16. At Week 28, participants were re-randomized to continue on ustekinumab (Treatment group B1) at Weeks 28 and 40.
Arm/Group | Through Week 28: ABP 654 | Through Week 28: Ustekinumab | Post Week 28: ABP 654 / ABP 654 | Post Week 28: Ustekinumab / ABP654 | Post Week 28: Ustekinumab / Ustekinumab | Post Week 28: ABP 654 Dose Intensification | Post Week 28: Ustekinumab Dose Intensification
All-Cause Mortality (participants affected / at risk) | 0/280 | 1/282 | 0/247 | 0/117 | 0/116 | 0/25 | 0/34
Serious Adverse Events (participants affected / at risk) | 7/280 | 5/282 | 1/247 | 1/117 | 3/116 | 1/25 | 0/34
Other Adverse Events (participants affected / at risk) | 21/280 | 15/282 | 36/247 | 22/117 | 17/116 | 9/25 | 2/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Through Week 28: ABP 654 (N=280) | Through Week 28: Ustekinumab (N=282) | Post Week 28: ABP 654 / ABP 654 (N=247) | Post Week 28: Ustekinumab / ABP654 (N=117) | Post Week 28: Ustekinumab / Ustekinumab (N=116) | Post Week 28: ABP 654 Dose Intensification (N=25) | Post Week 28: Ustekinumab Dose Intensification (N=34)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Through Week 28: ABP 654 (N=280) | Through Week 28: Ustekinumab (N=282) | Post Week 28: ABP 654 / ABP 654 (N=247) | Post Week 28: Ustekinumab / ABP654 (N=117) | Post Week 28: Ustekinumab / Ustekinumab (N=116) | Post Week 28: ABP 654 Dose Intensification (N=25) | Post Week 28: Ustekinumab Dose Intensification (N=34)
COVID-19 (Infections and infestations) | 6 | 4 | 23 | 15 | 10 | 5 | 1
Nasopharyngitis (Infections and infestations) | 7 | 3 | 9 | 1 | 7 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 7 | 6 | 6 | 3 | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 1 | 1 | 2 | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Due to non-convergence of the generalized linear model used for pre-specified analyses, ad hoc analyses were conducted for efficacy endpoints of PASI 75 response, PASI 100 response, and sPGA response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT04607980/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT04607980/SAP_001.pdf